CLINICAL TRIAL: NCT03277794
Title: Generating Evidence for a Comprehensive Support Package to Stabilize Youth Trajectories Out of Homelessness: A Tertiary Prevention Strategy
Brief Title: Generating Evidence for a Support Package to Stabilize Youth Trajectories Out of Homelessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/06/2017
Record Dates: First submitted 2017-08-14; First posted 2017-09-11 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Youth; Homelessness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional Case Management Only (Active Comparator): Participants in this arm will be provided with a transition-focused community support worker who will assist in areas ranging from general support and encouragement to assistance in navigating relevant systems. They will have weekly contacts with participants by phone, informal contact via text and email, and at least twice per month will visit the participant where they are residing. It is expected that all participants will engage a community support worker. The transitional case manager hired into this role will be highly experienced in case management for youth.
  Interventions: Behavioral: Transitional Case Management Only
- Full HOP-C Service (Experimental): Service provision will be provided by Loft and Covenant House for the transitional case management component, the peer component will be supported through Sketch Arts, and the mental health component will be provided by a post-doctoral fellow clinical psychologist and a mindfulness therapist from the Centre for Mindfulness Studies, supervised by Dr. Sean Kidd.
  Interventions: Behavioral: HOP-C

INTERVENTIONS:
Behavioral: HOP-C — Service provision will be provided by Loft and Covenant House for the transitional case management component, the peer component will be supported through Sketch Arts, and the mental health component will be provided by a post-doctoral fellow clinical psychologist and a mindfulness therapist from the Centre for Mindfulness Studies, supervised by Dr. Sean Kidd.
  Arms: Full HOP-C Service
Behavioral: Transitional Case Management Only — Participants in this arm will be provided with a transition-focused community support worker who will assist in areas ranging from general support and encouragement to assistance in navigating relevant systems. They will have weekly contacts with participants by phone, informal contact via text and email, and at least twice per month will visit the participant where they are residing. It is expected that all participants will engage a community support worker. The transitional case manager hired into this role will be highly experienced in case management for youth.
  Arms: Transitional Case Management Only

SUMMARY:
This project builds upon initial proof of concept work examining the optimal set of supports for youth who have recently exited homelessness - an intervention comprised of mental health and peer supports alongside transitional case management. This collaborative model will be tested as a proof-of-concept in Thunder Bay with Indigenous youth and a trial will be conducted in Toronto to optimize and determine the effectiveness of the existing model of support.

DETAILED DESCRIPTION:
In response to the challenges outlined above, and with the support of a grant from the Ontario Ministry of Child and Youth Services, the investigators developed and tested a tertiary prevention strategy called the Housing Outreach Program Collaborative (HOP-C) which launched in the summer of 2015. In this approach the investigators focused on collaborations and interventions that have the greatest potential to be effective with this population. The investigators brought together partners from a number of sectors in the GTA and have tested a 3-pronged set of supports (intervention described in detail in the methods):

* Transitional Case Management
* Mental Health Interventions: Group, individual, family
* Peer Support This is an intensive, 6-month critical time intervention - one that jointly addresses many points of vulnerability (mental health crises, housing instability, justice involvement) while fostering resilience and connection with resources in employment, education and training domains. It is unique in both content comprehensiveness and integrated process of delivery. Also important was the development of a collaborative and responsive partnering process, to facilitate effective organizational interfaces and seamless service integration so participants can experience a tailored and coherent set of supports. With CAMH, the Centre for Mindfulness Studies, Covenant House, LOFT, and SKETCH at the service level and the Wellesley Institute leading evaluation, the investigators have carefully attended to a collective impact framework.

This initiative has proven feasible and is demonstrating good outcomes - with excellent youth engagement, reports of lower social isolation, improved mental health, and engagement with resources, and spin-off benefits of closer collaboration between organizations. The investigators successfully met the target of youth engagement, with a total of 31 youth participating, minimal attrition (n=2), and the investigators observed no indications that HOP-C resulted in risk of any form, both with respect to the intervention itself and the mixed methods research methodology. This promising feasibility work formed the foundation from which the investigators were successful in obtaining a grant from the Local Poverty Reduction Fund to support the study described in this proposal.

Current Project Determine through a randomized trial in Toronto if the positive outcomes the investigators are observing are due solely or primarily to transitional case management and if the additional peer and mental health components are necessary.

Engaging in intensive, tertiary prevention shows clear promise in disrupting a cycle of poverty and marginalization at a critical time - if proven and scaled a key driver of chronic homelessness would be addressed.

Research Questions The objective of this two-part project is to examine the effectiveness and transferability of the Housing Outreach Program-Collaboration (HOP-C) transitional intervention. HOP-C has proven to be feasible with promising outcomes in the Toronto proof-of-concept work currently underway.

1. Are the benefits of the complex HOP-C intervention with all components in place greater than transitional case management in isolation?

• It is hypothesized that the full model will provide benefit in domains of housing stability, mental health, and quality of life that are significantly greater than case management alone.

The investigators have data in hand from their recent national work in the area which provides data on 'treatment as usual' or the outcomes that attend typically available supports. The proposed trial will unpack benefit and be essential in economic and viability arguments to be made going forward.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 16 and 26
* have obtained secure housing in a time period up to 12 months previously

Exclusion Criteria:

* none

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean A Kidd, Phd, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altena AM, Brilleslijper-Kater SN, Wolf JL. Effective interventions for homeless youth: a systematic review. Am J Prev Med. 2010 Jun;38(6):637-45. doi: 10.1016/j.amepre.2010.02.017. PMID 20494240
- [Background] Barber CC, Fonagy P, Fultz J, Simulinas M, Yates M. Homeless near a thousand homes: outcomes of homeless youth in a crisis shelter. Am J Orthopsychiatry. 2005 Jul;75(3):347-55. doi: 10.1037/0002-9432.75.3.347. PMID 16060731
- [Background] Boyatzis, R. E. (1998). Transforming Qualitative Information: Thematic Analysis and code Development. Thousand Oaks, California: Sage.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Bryman, A. (2006). Integrating quantitative and qualitative research: How is it done? Qualitative Research, 6, 97-113.
- [Background] Cloitre M, Courtois CA, Charuvastra A, Carapezza R, Stolbach BC, Green BL. Treatment of complex PTSD: results of the ISTSS expert clinician survey on best practices. J Trauma Stress. 2011 Dec;24(6):615-27. doi: 10.1002/jts.20697. Epub 2011 Dec 6. PMID 22147449
- [Background] Craig TK, Hodson S. Homeless youth in London: I. Childhood antecedents and psychiatric disorder. Psychol Med. 1998 Nov;28(6):1379-88. doi: 10.1017/s0033291798007351. PMID 9854279
- [Background] Research design: qualitative, quantitative and mixed methods approaches Research design: qualitative, quantitative and mixed methods approaches Creswell John W Sage 320 pound29 0761924426 0761924426 [Formula: see text]. Nurse Res. 2004 Sep 1;12(1):82-83. doi: 10.7748/nr.12.1.82.s2. PMID 28718745
- [Background] Frederick, T., Chwalek, M., Hughes, J., Karabanow, J., & Kidd, S.A. (2014). How stable is stable? Defining and measuring housing stability. Journal of Community Psychology, 42, 964-979*.
- [Background] Gaetz, S., Donaldson, J., Richter, T., & Gulliver, T. (2013). The State of Homelessness in Canada - 2013. Toronto: Canadian Homeless Research Network Press.
- [Background] Grabbe, L., Nguy, S. & Higgins, M. (2012). Spirituality development for homeless youth: A mindfulness meditation feasibility pilot. Journal of Child and Family Studies 21, 925-37.
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Hurn J, Kneebone I, Cropley M. Goal setting as an outcome measure: A systematic review. Clin Rehabil. 2006 Sep;20(9):756-72. doi: 10.1177/0269215506070793. PMID 17005500
- [Background] Hwang SW, Kirst MJ, Chiu S, Tolomiczenko G, Kiss A, Cowan L, Levinson W. Multidimensional social support and the health of homeless individuals. J Urban Health. 2009 Sep;86(5):791-803. doi: 10.1007/s11524-009-9388-x. Epub 2009 Jul 23. PMID 19629703
- [Background] Karabanow J. (2004). Being Young and Homeless: Understanding how youth enter and exit street life. New York, NY. Peter Lang Publishing INC.
- [Background] Karabanow, J., Hopkins, S., Kisely, S., Parker, J., Hughes, J., Gahagan, J., and Campbell, LA. (2007). Can You Be healthy on the Street?: Exploring the Health Experiences of Halifax Street Youth. The Canadian Journal of Urban Research, 16, 12-32.
- [Background] Karabanow, J. (2008). Getting off the Street: Exploring Young People's Street Exits. American Behavioral Scientist, 51, 772-788.
- [Background] Kerrigan D, Johnson K, Stewart M, Magyari T, Hutton N, Ellen JM, Sibinga EM. Perceptions, experiences, and shifts in perspective occurring among urban youth participating in a mindfulness-based stress reduction program. Complement Ther Clin Pract. 2011 May;17(2):96-101. doi: 10.1016/j.ctcp.2010.08.003. Epub 2010 Sep 16. PMID 21457899
- [Background] Kidd SA, Scrimenti K. Evaluating child and youth homelessness. Eval Rev. 2004 Aug;28(4):325-41. doi: 10.1177/0193841X04264820. PMID 15245623
- [Background] Kidd, S.A. (2006). Factors precipitating suicidality among homeless youth: A quantitative follow-up. Youth & Society, 37, 393-422.
- [Background] Kidd, S.A., & Davidson, L. (2007). "You have to adapt because you have no other choice.": The stories of strength and resilience of 208 homeless youth in New York City and Toronto. Journal of Community Psychology, 35, 219-238.
- [Background] Kidd S. Invited commentary: seeking a coherent strategy in our response to homeless and street-involved youth: a historical review and suggested future directions. J Youth Adolesc. 2012 May;41(5):533-43. doi: 10.1007/s10964-012-9743-1. PMID 22302217
- [Background] Kidd, S.A., Frederick, T., Karabanow, J.,Hughes, J., & Barbic, S. (2016). A mixed methods of recently homeless youth efforts to sustain housing and stability. Child and Adolescent Social Work Journal, 33, 207-218.
- [Background] Linehan, M. (2014). DBT Skills Training Manual Second Edition. New York: The Guilford Press.
- [Background] Milburn NG, Rice E, Rotheram-Borus MJ, Mallett S, Rosenthal D, Batterham P, May SJ, Witkin A, Duan N. Adolescents Exiting Homelessness Over Two Years: The Risk Amplification and Abatement Model. J Res Adolesc. 2009 Dec 1;19(4):762-785. doi: 10.1111/j.1532-7795.2009.00610.x. PMID 25067896
- [Background] Public Health Agency of Canada. (2006). Street Youth in Canada. www.publichealth.gc.ca/sti
- [Background] Rew L, Horner SD. Personal strengths of homeless adolescents living in a high-risk environment. ANS Adv Nurs Sci. 2003 Apr-Jun;26(2):90-101. doi: 10.1097/00012272-200304000-00002. PMID 12795538
- [Background] Rosenthal D, Rotheram-Borus MJ, Batterham P, Mallett S, Rice E, Milburn NG. Housing stability over two years and HIV risk among newly homeless youth. AIDS Behav. 2007 Nov;11(6):831-41. doi: 10.1007/s10461-007-9235-6. Epub 2007 May 12. PMID 17497219
- [Background] Roy E, Haley N, Leclerc P, Sochanski B, Boudreau JF, Boivin JF. Mortality in a cohort of street youth in Montreal. JAMA. 2004 Aug 4;292(5):569-74. doi: 10.1001/jama.292.5.569. PMID 15292082
- [Background] Roy E, Haley N, Boudreau JF, Leclerc P, Boivin JF. The challenge of understanding mortality changes among street youth. J Urban Health. 2010 Jan;87(1):95-101. doi: 10.1007/s11524-009-9397-9. Epub 2009 Dec 29. PMID 20039140
- [Background] Roy E, Robert M, Fournier L, Vaillancourt E, Vandermeerschen J, Boivin JF. Residential trajectories of street youth-the Montreal Cohort Study. J Urban Health. 2014 Oct;91(5):1019-31. doi: 10.1007/s11524-013-9860-5. PMID 24515932
- [Background] Rush B, Castel S, Brands B, Toneatto T, Veldhuizen S. Validation and comparison of diagnostic accuracy of four screening tools for mental disorders in people seeking treatment for substance use disorders. J Subst Abuse Treat. 2013 Apr;44(4):375-83. doi: 10.1016/j.jsat.2012.08.221. Epub 2012 Oct 23. PMID 23098381
- [Background] Sandelowski M. Sample size in qualitative research. Res Nurs Health. 1995 Apr;18(2):179-83. doi: 10.1002/nur.4770180211. PMID 7899572
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Slesnick N, Kang MJ, Bonomi AE, Prestopnik JL. Six- and twelve-month outcomes among homeless youth accessing therapy and case management services through an urban drop-in center. Health Serv Res. 2008 Feb;43(1 Pt 1):211-29. doi: 10.1111/j.1475-6773.2007.00755.x. PMID 18211526
- [Background] Slesnick N, Bartle-Haring S, Dashora P, Kang MJ, Aukward E. Predictors of Homelessness Among Street Living Youth. J Youth Adolesc. 2008;37(4):465-474. doi: 10.1007/s10964-007-9188-0. PMID 18584069
- [Background] Slesnick N, Dashora P, Letcher A, Erdem G, Serovich J. A Review of Services and Interventions for Runaway and Homeless Youth: Moving Forward. Child Youth Serv Rev. 2009 Jul;31(7):732-742. doi: 10.1016/j.childyouth.2009.01.006. PMID 20161294
- [Background] Snyder CR, Harris C, Anderson JR, Holleran SA, Irving LM, Sigmon ST, Yoshinobu L, Gibb J, Langelle C, Harney P. The will and the ways: development and validation of an individual-differences measure of hope. J Pers Soc Psychol. 1991 Apr;60(4):570-85. doi: 10.1037//0022-3514.60.4.570. PMID 2037968
- [Background] Stergiopoulos V, Gozdzik A, O'Campo P, Holtby AR, Jeyaratnam J, Tsemberis S. Housing First: exploring participants' early support needs. BMC Health Serv Res. 2014 Apr 13;14:167. doi: 10.1186/1472-6963-14-167. PMID 24725374
- [Background] Tevendale HD, Comulada WS, Lightfoot MA. Finding shelter: two-year housing trajectories among homeless youth. J Adolesc Health. 2011 Dec;49(6):615-20. doi: 10.1016/j.jadohealth.2011.04.021. PMID 22098772
- [Background] Unesco. (2014, July 4). Street Children. Retrieved from: http://www.unesco.org/new/en/social-and-human-sciences/themes/fight-against-discrimination/education-of-children-in-need/street-children/.
- [Background] Wagnild G.M. The Resilience Scale user's guide for the US English version of the Resilience Scale and the 14- Item Resilience Scale (RS-14). Worden, MT: The Resilience Center. 2010.
- [Background] Yalom, I.D. & Leszcz, M. (2005). The Theory & Practice of Group Psychotherapy, 5th ed. N.Y.: Basic Books.
- [Derived] Kidd SA, Vitopoulos N, Frederick T, Leon S, Wang W, Mushquash C, McKenzie K. Trialing the feasibility of a critical time intervention for youth transitioning out of homelessness. Am J Orthopsychiatry. 2020;90(5):535-545. doi: 10.1037/ort0000454. Epub 2020 Apr 20. PMID 32309974
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addictions teaching hospital. — http://www.camh.ca/en/research/Pages/research.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Transitional Case Management Only: Participants in this arm will be provided with a transition-focused community support worker who will assist in areas ranging from general support and encouragement to assistance in navigating relevant systems. They will have weekly contacts with participants by phone, informal contact via text and email, and at least twice per month will visit the participant where they are residing. It is expected that all participants will engage a community support worker. The transitional case manager hired into this role will be highly experienced in case management for youth.
  Transitional Case Management Only: Participants in this arm will be provided with a transition-focused community support worker who will assist in areas ranging from general support and encouragement to assistance in navigating relevant systems. They will have weekly contacts with participants by phone, informal contact via text and email, and at least twice per month will visit the participant where they are residing.
Period: Overall Study
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Started | 31 | 34
Completed | 28 | 30
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrew due to high acuity | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transitional Case Management Only: Transitional Case Management Only: Participants in this arm will be provided with a transition-focused community support worker who will assist in areas ranging from general support and encouragement to assistance in navigating relevant systems. They will have weekly contacts with participants by phone, informal contact via text and email, and at least twice per month will visit the participant where they are residing.
- Total: Total of all reporting groups
Arm/Group | Transitional Case Management Only | Full HOP-C Service | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.74 (2.03) | 21.76 (2.14) | 21.75 (2.07)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Other | 17 | 22 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - North American | 5 | 5 | 10
  Black - African | 5 | 3 | 8
  Black - Caribbean | 3 | 4 | 7
  Mixed Heritage | 2 | 4 | 6
  Other/Not Specified | 16 | 18 | 34
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 21 | 22 | 43
  Bi-Sexual | 3 | 4 | 7
  Prefer not to answer | 2 | 2 | 4
  Other/Not Specified | 5 | 6 | 11
Highest Education [Count of Participants; unit: Participants]
  Some High School | 14 | 7 | 21
  Completed High School | 7 | 11 | 18
  Transitional Program | 6 | 11 | 17
  Other/Not Specified | 4 | 5 | 9
Homelessness - Lifetime Length [Count of Participants; unit: Participants]
  6-12 Months | 7 | 11 | 18
  1-2 years | 10 | 6 | 16
  2-3 years | 1 | 10 | 11
  3+ years | 13 | 7 | 20
NEET - Not in Employment, Education or Training [Count of Participants; unit: Participants] | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Housing
Description: Participants coded in a binary manner as having gained or sustained housing (binary positive) or lost (binary negative) based on assessment of the participant's trajectory from baseline to 6 months.
Time Frame: Change from Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
Participants | 25 | 28
Statistical Analysis 1: Comparison: Transitional Case Management Only vs Full HOP-C Service; Full HOP-C Service (Treatment) vs. Transitional Case Management Only (Control); Test type: Other; p = 0.354, Regression, Logistic; Odds Ratio (OR) = 2.28, Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Transitional Case Management Only vs Full HOP-C Service; Full HOP-C Service (Treatment) vs. Transitional Case Management Only (Control); Test type: Other; p = 0.465, Regression, Logistic; Odds Ratio (OR) = 2.01, Standard Error of Mean 0.95

2. Primary Outcome: Employment/Education
Description: Participants coded in a binary manner as having gained or sustained education or employment (binary positive) or lost (binary negative) based on assessment of the participant's trajectory from baseline to 6 months.
Time Frame: Change from baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
Participants | 18 | 24
Statistical Analysis 1: Comparison: Transitional Case Management Only vs Full HOP-C Service; Full HOP-C Service (Treatment) vs. Transitional Case Management Only (Control); Test type: Other; p = 0.159, Regression, Logistic; Odds Ratio (OR) = 2.31, Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Transitional Case Management Only vs Full HOP-C Service; Full HOP-C Service (Treatment) vs. Transitional Case Management Only (Control); Test type: Other; p = 0.200, Regression, Linear; Odds Ratio (OR) = 2.30, Standard Error of Mean 0.64

3. Primary Outcome: Mental Health
Description: Participants coded in a binary manner as having gained or sustained mental health status without crises (binary positive) or experienced a crises that impacted major life domains (binary negative) based on assessment of the participant's trajectory from baseline to 6 months.
Time Frame: Change from baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
Participants | 20 | 27
Statistical Analysis 1: Comparison: Transitional Case Management Only vs Full HOP-C Service; Full HOP-C Service (Treatment) vs. Transitional Case Management Only (Control); Test type: Other; p = 0.121, Regression, Logistic; Odds Ratio (OR) = 3.18, Standard Error of Mean 0.74
Statistical Analysis 2: Comparison: Transitional Case Management Only vs Full HOP-C Service; Full HOP-C Service (Treatment) vs. Transitional Case Management Only (Control); Test type: Other; p = 0.134, Regression, Logistic; Odds Ratio (OR) = 3.63, Standard Error of Mean 0.85

4. Primary Outcome: Housing Security Scale
Description: The Housing Security Scale contains 12 items on a 5 point likert scale (Frederick et al., 2014). Scores range from "strongly disagree" (minimum = 1) to "strongly agree" (maximum = 5). Higher scores indicate better outcomes. Mean item range is 1-5 with pre-post difference reported.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | 0.017 (0.129) | 0.153 (0.098)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.899, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.128, Regression, Linear — Unadjusted

5. Primary Outcome: Housing Security Scale (Subjective Housing Stability Subscale)
Description: The Housing Security Scale contains a 4 item subscale that measures subjective housing satisfaction and perception of housing stability (Frederick et al., 2014). Scores range from "strongly disagree" (minimum = 1) to "strongly agree" (maximum = 5). Higher scores indicate better outcomes with a mean range of 1-5 with pre-post change reported.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | -0.259 (0.196) | 0.422 (0.167)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.198, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.017, Regression, Linear — Unadjusted

6. Secondary Outcome: Mental Health Continuum - Short Form
Description: Mental Health Continuum - Short Form assess mental health and addictions by measuring emotional, psychological and social well-being. It contains 14 items on a 6 point scale ranging from at minimum "never" (0) to, at maximum, "every day" (5). Higher scores indicate better outcomes. Range is 0-5 (means) with pre-post differences reported.
Time Frame: Change from baseline to 6 month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | 0.276 (0.157) | 0.077 (0.141)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.091, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.591, Regression, Linear — Unadjusted

7. Secondary Outcome: Cognitive and Affective Mindfulness Scale
Description: Cognitive and Affective Mindfulness Scale Revised was used to measure mindfulness and has demonstrated acceptable reliability (Feldman, Hayes, Kumar, Greeson, & Laurenceau, 2007). It contains 10 items. The minimum score is "rarely/Not at all" (1) and the maximum score is "almost always" (4). Higher scores indicate better outcomes with a mean item range from 1-4 with pre-post mean change reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | 0.226 (0.099) | 0.176 (0.058)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.030, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.005, Regression, Linear — Unadjusted

8. Secondary Outcome: Community Integration Scale
Description: Behavioural and psychological aspects of community integration was examined using Community Integration Scale The scale contains 7 dichotomous questions with higher scores indicating greater community integration (better outcomes). Mean item range is 0-1 with mean change reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | -0.108 (0.075) | 0.008 (0.045)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.163, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.865, Regression, Linear — Unadjusted

9. Secondary Outcome: Community Integration Measure
Description: Behavioural and psychological aspects of community integration were examined using the Community Integration Measure. The measure contains 6 items scored on a 5 point scale ranging from, at minimum, "always disagree" (1) to, at maximum, "always agree" (5). Higher scores indicating better outcomes with an item mean range from 1-5 with mean pre-post differences reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | -0.006 (0.239) | -0.051 (0.163)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.980, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.758, Regression, Linear — Unadjusted

10. Secondary Outcome: Resilience Scale
Description: Resilience will be measured using the 10-item Resilience Scale. Each item score ranges from, at minimum, "Not true at all" (0) to, at maximum, "True nearly all the time" (4) with higher scores indicating better outcomes. Mean item range is from 0-4 with pre-post change in means reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | 0.252 (0.159) | 0.093 (0.065)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.124, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.168, Regression, Linear — Unadjusted

11. Secondary Outcome: Adults Hope Scale
Description: Adult Hope Scale, a cognitive measure of hope, was employed. This self-report questionnaire contains 8 questions that are each scored on an 8 point Likert scale with scores ranging from "Definitely False" to "Definitely True". Higher scores indicate better outcomes. Mean item range is minimum 1 to maximum 8 with pre-post mean differences reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale | 0.218 (0.276) | -0.038 (0.099)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Test type: Other; p = 0.436, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Test type: Other; p = 0.706, Regression, Linear — Unadjusted

12. Secondary Outcome: GAIN Short Screener (CAMH Modified)
Description: Mental health (and addictions) was measured using the Global Assessment of Individual Needs Short Screener, which includes 22 items scored on a 5 point scale ranging from "never" (0) as the minimum score and "past month" (4) as the maximum score. Higher scores indicate worse outcomes. Mean item range is 0-4 with pre-post mean change reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale
  Internalizing | -0.124 (0.236) | -0.265 (0.191)
  Externalizing | -0.151 (0.15) | -0.212 (0.171)
  Substance Use | -0.308 (0.184) | -0.291 (0.147)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Internalizing; Test type: Other; p = 0.604, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Internalizing; Test type: Other; p = 0.177, Regression, Linear — Unadjusted
Statistical Analysis 3: Comparison: Transitional Case Management Only; Externalizing; Test type: Other; p = 0.325, Regression, Linear — Unadjusted
Statistical Analysis 4: Comparison: Full HOP-C Service; Externalizing; Test type: Other; p = 0.227, Regression, Linear — Unadjusted
Statistical Analysis 5: Comparison: Transitional Case Management Only; Substance Use; Test type: Other; p = 0.106, Regression, Linear — Unadjusted
Statistical Analysis 6: Comparison: Full HOP-C Service; Substance Use; Test type: Other; p = 0.058, Regression, Linear — Unadjusted

13. Secondary Outcome: Medical Outcomes Study (MOS) Social Support Survey
Description: We used a modified version of the Medical Outcomes Study Social Support Survey to measure social support. It is a 15-item 5-point Likert-type scale. The maximum score is "all of the time" (5) and the minimum score is "none of the time" (1). Higher score indicates better outcome. Item mean range is 1-5 with pre-post mean difference reported.
Time Frame: Change from baseline to 6 month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale
  Emotional Supports | 0.043 (0.247) | 0.174 (0.196)
  Tangible Supports | 0.110 (0.264) | -0.003 (0.194)
  Affectionate Supports | -0.115 (0.297) | 0.333 (0.227)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Emotional Supports; Test type: Other; p = 0.862, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Emotional Supports; Test type: Other; p = 0.382, Regression, Linear — Unadjusted
Statistical Analysis 3: Comparison: Transitional Case Management Only; Tangible Supports; Test type: Other; p = 0.680, Regression, Linear — Unadjusted
Statistical Analysis 4: Comparison: Full HOP-C Service; Tangible Supports; Test type: Other; p = 0.988, Regression, Linear — Unadjusted
Statistical Analysis 5: Comparison: Transitional Case Management Only; Affectionate; Test type: Other; p = 0.701, Regression, Linear — Unadjusted
Statistical Analysis 6: Comparison: Full HOP-C Service; Affectionate; Test type: Other; p = 0.154, Regression, Linear — Unadjusted

14. Secondary Outcome: World Health Organization Quality of Life Scale - BREF
Description: The brief World Health Organization Quality of Life Scale - BREF contains 26 items, each scored from 1 to 5 with various labels for each score (e.g. 1= "very poor" for item 1 and 1= "very dissatisfied" for item 2). Higher scores indicate better outcomes with a mean item range of 1-5 with pre-post mean change reported.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transitional Case Management Only | Full HOP-C Service
Number analyzed (Participants) | 28 | 30
score on a scale
  Physical Health | 0.201 (0.552) | 0.717 (0.484)
  Psychological | -0.117 (0.432) | 0.086 (0.355)
  Social | 0.308 (0.869) | 0.099 (0.376)
  Environment | 0.124 (0.596) | 0.843 (0.407)
Statistical Analysis 1: Comparison: Transitional Case Management Only; Physical Health; Test type: Other; p = 0.719, Regression, Linear — Unadjusted
Statistical Analysis 2: Comparison: Full HOP-C Service; Physical Health; Test type: Other; p = 0.150, Regression, Linear — Unadjusted
Statistical Analysis 3: Comparison: Transitional Case Management Only; Psychological; Test type: Other; p = 0.789, Regression, Linear — Unadjusted
Statistical Analysis 4: Comparison: Full HOP-C Service; Psychological; Test type: Other; p = 0.811, Regression, Linear — Unadjusted
Statistical Analysis 5: Comparison: Transitional Case Management Only; Social; Test type: Other; p = 0.726, Regression, Linear — Unadjusted
Statistical Analysis 6: Comparison: Full HOP-C Service; Social; Test type: Other; p = 0.795, Regression, Linear — Unadjusted
Statistical Analysis 7: Comparison: Transitional Case Management Only; Environment; Test type: Other; p = 0.837, Regression, Linear — Unadjusted
Statistical Analysis 8: Comparison: Full HOP-C Service; Environment; Test type: Other; p = 0.048, Regression, Linear — Unadjusted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Transitional Case Management Only | Full HOP-C Service
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/34
Other Adverse Events (participants affected / at risk) | 0/31 | 0/34

LIMITATIONS AND CAVEATS:
Variability in youth service need resulting in variable effectiveness of treatment. In attempt to normalize the control group, it became less generalizable. RCT challenges with engagement and trust.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03277794/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT03277794/ICF_001.pdf